CLINICAL TRIAL: NCT06014060
Title: 24 Versus 12-Month Dual Antiplatelet Therapy After Drug-Eluting Stent in Patients With Elevated Lipoprotein(a) Levels: A Prospective, Multicenter, Double-Blind, Placebo-Controlled Randomized Trial
Acronym: DAPT-Lp(a)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Kefei Dou, MD, Professor, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Lipoprotein(a) and prognosis
Record Dates: First submitted 2023-08-23; First posted 2023-08-28 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Elevated Lipoprotein(a) Level; Coronary Artery Disease; Drug-Eluting Stent; Dual Antiplatelet Therapy
Keywords: Lipoprotein(a); Coronary Artery Disease; Drug-Eluting Stent; Percutaneous Coronary Intervention; Dual Antiplatelet Therapy
MeSH Terms: conditions — Coronary Artery Disease | interventions — 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study investigators, clinicians, participants, clinical assessors (including the follow-up research personnel, clinical events committee [CEC]) were unaware of the study-group assignments. All potential events were adjudicated according to prespecified criteria by an independent clinical events committee whose members were unaware of the trial-group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 24 Months DAPT (Experimental): Dual antiplatelet therapy consisting of aspirin and clopidogrel will be continued for 12 months after randomisation.
  Interventions: Procedure: 24 Months DAPT
- 12 Months DAPT (Active Comparator): Aspirin + a placebo that is exactly the same in size, color, smell, taste and appearance as clopidogrel were administered for 12 months after randomisation.
  Interventions: Procedure: 12 Months DAPT

INTERVENTIONS:
Procedure: 24 Months DAPT — All subjects will receive co-administration of aspirin (100 mg/day) and clopidogrel (75 mg/day) for 12 months after randomization. The DAPT will last for 24 months after PCI.
  Arms: 24 Months DAPT
Procedure: 12 Months DAPT — All the subjects will receive aspirin (100 mg/day) + a placebo that is exactly the same in size, color, smell, taste and appearance as clopidogrel for 12 months after randomization. The DAPT will last for 12 months after PCI.
  Arms: 12 Months DAPT

SUMMARY:
1. Main objective Among patients with elevated Lp(a) levels (>30mg/dL) who did not experience cardiovascular events or BARC type 2, 3, or 5 bleeding within 12 months after PCI and DES implantation, was it possible to reduce the primary adverse cardiovascular and cerebrovascular events (a composite endpoint consisting of all-cause death, non-fatal myocardial infarction, and stroke) by extending the duration of DAPT (24 months) compared to the standard duration (12 months)? (Efficacy test)
2. Secondary Objectives Key secondary research objective: Among patients with elevated Lp(a) levels (> 30mg/dL) who underwent PCI and received DES implantation within 12 months after the procedure, and who did not experience cardiovascular events or BARC type 2, 3, or 5 bleeding, whether extending the DAPT duration (24 months) compared to the standard DAPT duration (12 months) does not result in an increase in clinical net adverse events (a composite endpoint consisting of all-cause death, non-fatal myocardial infarction, stroke, and BARC type 3 or 5 bleeding) compared to the standard DAPT duration. (Non-inferiority test) Other secondary research objectives: To evaluate the differences in the incidence of the composite endpoint consisting of BARC type 3 or 5 bleeding (the primary safety endpoint) between extending the DAPT duration (24 months) and the standard DAPT duration (12 months); the differences in the incidence of the composite endpoint consisting of cardiovascular death and myocardial infarction; the differences in the incidence of the composite endpoint consisting of all-cause death and myocardial infarction; the differences in the incidence of stent thrombosis; the differences in the incidence of any myocardial infarction; the differences in the incidence of target vessel myocardial infarction; the differences in the incidence of stroke; the differences in the incidence of ischemic stroke; the differences in the incidence of hemorrhagic stroke; the differences in the incidence of cardiovascular death; the differences in the incidence of all-cause death; the differences in the incidence of repeat revascularization; the differences in the incidence of target vessel revascularization; the differences in the incidence of BARC type 2, 3, or 5 bleeding; the differences in the incidence of any bleeding.

DETAILED DESCRIPTION:
Lp(a) levels play an important role in predicting subsequent ischemic events in patients with established coronary artery disease (CAD), especially those who underwent PCI. However, there are still no approved pharmacologic therapies that specifically target high Lp(a) levels.

DAPT consisting of aspirin and a P2Y12 receptor inhibitor represents the cornerstone of pharmacological treatment aimed at preventing thrombotic complications after PCI. Considering that Lp(a) has a prothrombotic effect through its inactive, plasminogen-like protease domain on apo(a), the investigators speculate that prolonged DAPT may have a beneficial effect on reducing future ischemic events in patients with elevated Lp(a) levels after PCI. Some observational studies revealed that DAPT > 1 year was significantly associated with lower risk of cardiovascular events compared with DAPT ≤ 1 year in patients with elevated Lp(a) levels who were event-free at 1 year after PCI with DES. However, the relative efficacy and safety of prolonged DAPT versus standard DAPT in this high-risk population has never been assessed in randomized controlled trials (RCTs).

The DAPT-Lp(a) trial is a multicenter, parallel-group, randomized controlled trial with blinded end-point evaluation. Consecutive patients with Lp(a) levels>30mg/dL who meet the inclusion criteria and none of the exclusion criteria will be randomized in a 1:1 fashion to 24-month DAPT group or 12-month DAPT group. The investigators hypothesise that, in patients with Lp(a) levels >30mg/dL who were event-free at 1 year after PCI with DES, 24-month DAPT is superior to 12-month DAPT with respect to major adverse cardiovascular and cerebrovascular events (primary end point), while it is non-inferior to 12-month DAPT with respect to net adverse clinical events (key secondary end point).

The investigators estimated that 3,300 patients would be needed to provide the necessary number of confirmed endpoints to test the study hypothesis. Patients will be followed up at 3, 6, 9, 12 months after randomization. All analyses will be performed according to the intention-to-treat (ITT) principle.

ELIGIBILITY:
Inclusion Criteria:

1. Male or nonpregnant female between 18-75 years;
2. Subjects with Lp(a) levels > 30mg/dL before percutaneous coronary intervention (PCI);
3. PCI procedure with drug-eluting stent (DES) implantation and no cardiovascular events or BARC type 2, 3, or 5 bleeding events occurring within 12 months after the procedure
4. Subjects (or legal guardian) understand the trial requirements and the treatment procedures and provides written informed;

Exclusion Criteria:

1. Subjects with Lp(a) < 30mg/dL or Lp(a) level unavailable before PCI;
2. Subjects who experience adverse cardiovascular events (death, myocardial infarction, stent thrombosis, stroke, repeat coronary revascularization, or Bleeding Academic Research Consortium [BARC] type 2, 3 or 5 bleeding) within 1-year after PCI;
3. BARC type 2, 3, or 5 bleeding occurred before PCI
4. Unable to tolerate DAPT therapy or anticoagulant therapy at the same time, long-term use of non-steroidal anti-inflammatory drugs is required Or glucocorticoids;
5. Discontinuation of DAPT for ≥14 days for planned surgical procedures in the next 12 months;
6. Systolic blood pressure < 90mmHg for > 30 minutes accompanied by hypoperfusion symptoms or systolic blood pressure ≥ 90mmHg is maintained with mechanical/pharmacologic hemodynamic support;
7. Persistent symptoms of myocardial ischemia;
8. Moderate to severe heart failure (New York Heart Association [NYHA] Functional Classification III or IV) or last known left ventricular ejection fraction (LVEF) < 40%;
9. Severe valvular heart disease, myocarditis or cardiomyopathy;
10. Severe hepatic insufficiency (ALT or AST > 3 times upper limit of normal, total bilirubin > 2.5 times upper limit of normal);
11. Severe renal dysfunction, defined as creatinine clearance <30 mL/min or estimated glomerular filtration (eGFR) rate less than 30 ml/min/1.73m2, or requirement for peritoneal dialysis or hemodialysis for renal insufficiency;
12. Severe acute or chronic infectious disease;
13. History of severe rheumatic immune disease or malignant tumor;
14. Currently receiving treatment in another investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study(ies), or receiving other investigational agent(s);
15. Drug or alcohol abuse, and inability/unwillingness to abstain from drug abuse and excessive alcohol consumption during the study;
16. Recipient of any major organ transplant (eg, lung, liver, heart, bone marrow, renal);
17. Known significant active and uncontrolled disease, or any medical, physical condition, as judged by the investigator Or surgical status, may interfere with participation in this study
18. Mental/psychological disorder or any other reason that the subject is expected to have difficulty complying with the study requirements or understanding the participants With the objectives and potential risks of the study;
19. To the knowledge of the investigator, subjects were unlikely to follow up or were not expected to complete 1 year of follow-up;
20. Life expectancy is less than 1 year;

22. Refusal to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3300 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular and cerebrovascular event (MACCE) | 12 months after randomization
  The primary endpoint was major adverse cardiovascular and cerebrovascular event (MACCE), defined as a composite of all-cause death, non-fatal myocardial infarction or stroke.
BARC type 3 or 5 bleeding | 12 months after randomization
  Number of patients with a first occurrence of adjudicated BARC type 3 or 5 bleeding

SECONDARY OUTCOMES:
Net adverse clinical event (NACE) | 12 months after randomization
  The key secondary endpoint was net adverse clinical event, defined as a composite of all-cause death, non-fatal myocardial infarction, stroke or Bleeding Academic Research Consortium (BARC)] type 3 or 5 bleeding.
Cardiovascular death or myocardial infarction | 12 months after randomization
  Number of patients with a first occurrence of adjudicated composite of cardiovascular death or myocardial infarction.
All-cause death or myocardial infarction | 12 months after randomization
  Number of patients with a first occurrence of adjudicated composite of all-cause death or myocardial infarction.
Stent thrombosis | 12 months after randomization
  Number of patients with the adjudicated stent thrombosis.
Any myocardial infarction | 12 months after randomization
  Number of patients with a first occurrence of adjudicated any myocardial infarction.
Target vessel myocardial infarction | 12 months after randomization
  Number of patients with a first occurrence of adjudicated target vessel myocardial infarction.
Stroke | 12 months after randomization
  Number of patients with a first occurrence of adjudicated stroke.
Ischemic stroke | 12 months after randomization
  Number of patients with a first occurrence of adjudicated ischemic stroke.
Hemorrhagic stroke | 12 months after randomization
  Number of patients with a first occurrence of adjudicated hemorrhagic stroke.
Cardiovascular death | 12 months after randomization
  Number of patients with the occurrence of adjudicated cardiovascular death.
All-cause death | 12 months after randomization
  Number of patients with a first occurrence of adjudicated confirmed all-cause death
Repeat revascularization | 12 months after randomization
  Number of patients with a first occurrence of adjudicated repeat revascularization.
Target vessel revascularization | 12 months after randomization
  Number of patients with a first occurrence of adjudicated target vessel revascularization.
BARC type 2, 3 or 5 bleeding | 12 months after randomization
  Number of patients with a first occurrence of adjudicated BARC type 2, 3 or 5 bleeding.
Any bleeding | 12 months after randomization
  Number of patients with a first occurrence of adjudicated any bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Kefei Dou, MD, PhD, Principal Investigator — Fuwai Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College; Kongyong Cui, MD, PhD, Principal Investigator — Fuwai Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No